CLINICAL TRIAL: NCT00660088
Title: Tolerability, Safety, And Pharmacokinetics Of Three Formulations Of Oral Ketasyn™ (Ac-1202) Administered For Fourteen Days, With Or Without Titration, In Healthy Elderly Volunteers
Brief Title: Safety of Three Formulations of Ketasyn Administered for 14 Days in Healthy Elderly
Status: Completed | Type: Observational
Sponsor: Cerecin (Industry)
Responsible Party: Lauren Costantini, PhD; Vice President Clinical Development, Accera, Inc.
Other Study IDs: KET-08-004
Record Dates: First submitted 2008-04-11; First posted 2008-04-17 (Estimated); Last update posted 2008-10-08 (Estimated); Status verified 2008-10

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — plasma beta-hydroxybutyrate
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- 1: 10 gram x 7 days, then 20 gram x 7 days active ingredient of original formulation
  Interventions: Other: Ketasyn
- 2: 20 grams x 14 days active ingredient of original formulation
  Interventions: Other: Ketasyn
- 3: 10 grams x 7 days; then 20 grams x 7 days of low protein formulation
  Interventions: Other: Ketasyn
- 4: 20 grams x 14 days of low protein formulation
  Interventions: Other: Ketasyn
- 5: 10 grams x 7 days; then 20 grams x 7 days of high protein formulation
  Interventions: Other: Ketasyn
- 6: 20 grams x 14 days of high protein formulation
  Interventions: Other: Ketasyn

INTERVENTIONS:
Other: Ketasyn — 10g for 7 days, 20g for 7 or 14 days

SUMMARY:
AC-1202 (Ketasyn) is a nutritional beverage currently being studied in neurodegenerative conditions including Alzheimer's disease. The current study is a randomized, open-label trial to compare the safety, tolerability, and PK profiles of 3 formulations of Ketasyn administered on a daily basis for 14 days, with and without a 7-day titration period, in normal, healthy elderly volunteers.

DETAILED DESCRIPTION:
Sixty healthy, elderly volunteers between the ages of 55 and 85 will be enrolled at one of four clinical sites in the Tampa/St. Petersburg area. Subjects with a history of GI inflammatory conditions (e.g., IBS or diverticulitis) or other clinically significant abnormalities will be excluded from enrollment. Subjects will be randomized to one of two dosing regimens (with or without a 7-day titration period) and to one of three formulations of Ketasyn containing the identical amount of active ingredient, but different amounts of proteins and carbohydrates. Subjects assigned to Group 1 will receive 10 grams active ingredient daily on Days 1-7, followed by a daily dose of 20 grams active ingredient on Days 8-14. Subjects assigned to Group 2 will receive 20 grams active ingredient on Days 1-14. All subjects will have clinic visits on Day 1 and 14; subjects assigned to Group 1 will also have a clinic visit on Day 8. Subjects will fast prior to each clinic visit and have vital signs and routine lab tests performed prior to dosing. A standard breakfast will be served along with the study product, following which blood samples will be collected for product concentration levels.

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on physical exam, vital signs, medical history, ECG, or laboratory results

Exclusion Criteria:

* Type 1 or uncontrolled Type 2 diabetes
* History of or current inflammation of GI system, e.g. IBS, diverticular disease, gastric or duodenal ulcers, severe GERD requiring daily medication
* History (within past 60 days) of infections
* Clinically significant renal, hepatic, or hematologic abnormalities

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy elderly male and female subjects 55 - 85 years of age
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2008-04; Primary Completion 2008-06 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Plasma peak concentration levels and AUC | two weeks

SECONDARY OUTCOMES:
Incidence and severity of adverse events | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Lauren Costantini, PhD, Study Director — Cerecin
Locations (1):
- Meridien Research Center, St. Petersburg, Florida, United States